CLINICAL TRIAL: NCT02366754
Title: rTMS: A Treatment to Restore Function After Severe TBI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Edward Hines Jr. VA Hospital (U.S. Federal Agency)
Collaborators: Northwestern University (Other)
Responsible Party: Principal Investigator, Theresa Pape, Research Health Scientist, Edward Hines Jr. VA Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDMRP-PT130274
Record Dates: First submitted 2015-01-26; First posted 2015-02-19 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Traumatic Brain Injury
Keywords: Transcranial Magnetic Stimulation
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active rTMS (Experimental): The intervention consists of 30 active rTMS sessions. Each session is comprised of 300 trains of paired pulses with the following parameters: 100µs paired pulses separated by 100ms inter-pulse-intervals and a five second inter-train-interval. Pulse intensity will be set at 110% of each participant's motor threshold. Active rTMS sessions will be provided two times per day with a 70mm figure-of-eight coil over the left dorsolateral prefrontal cortex. Two Magstim-2002 units and a Bistim2 module will be used to administer active rTMS. Participants assigned to the active rTMS group will receive a total of 1.8 seconds of stimulation. Active rTMS will be administered 2 times daily with the following weekly schedule: 2 days of rTMS, 1 day of rest, 2 days of rTMS, 2 days of rest.
  Interventions: Device: rTMS
- Placebo rTMS (Sham Comparator): The intervention consists of 30 placebo rTMS sessions. Each session is comprised of 300 paired-pulse trains with the following parameters: 100µs paired pulses separated by 100ms inter-pulse-intervals and a five second inter-train-interval. Placebo rTMS sessions will be provided two times per day with a 70mm figure-of-eight coil over the left DLPFC. Two Magstim-2002 units and a Bistim2 module will be used to administer placebo rTMS. The placebo coil simulates magnetic stimulation, but does not actually emit a pulse. Participants assigned to the placebo rTMS group will receive 0 seconds of stimulation. Placebo rTMS will be administered with the following weekly schedule: 2 days of rTMS, 1 day of rest, 2 days of rTMS, 2 days of rest.
  Interventions: Device: Placebo rTMS

INTERVENTIONS:
Device: rTMS — Repetitive TMS is a non-invasive neural stimulation technique achieved via electromagnetic induction. An insulated metal coil is placed on the scalp and short discharges of electric current are directed through the coil producing a magnetic field. This magnetic field is accompanied by an electric field that passes through the skull inducing currents in the tissue beneath the coil. If a cell beneath the coil is viable, then rTMS initiates or inhibits an action potential affecting ongoing neural activity. 30 sessions of active rTMS are provided.
  Arms: Active rTMS
Device: Placebo rTMS — The placebo coil simulates magnetic stimulation, but does not actually emit a pulse. The placebo coil looks, sounds and feels like an active rTMS coil. The placebo coil, visually identical to the active coil, provides a slight sensory sensation and discharge noise (i.e., clicking) nearly identical to that of the active coil.
  Arms: Placebo rTMS

SUMMARY:
The purpose of this study is to address the need for targeted treatments that induce functional and structural changes in the brain, ultimately improving neurobehavioral functioning, the investigators propose examining the therapeutic effectiveness of repetitive Transcranial Magnetic Stimulation (rTMS). The objective is to improve functional recovery for persons remaining in vegetative (VS) and minimally conscious (MCS) states 3 to 24 months after severe TBI. The approach is to determine the neurobehavioral effect of rTMS, the relationship between neurobehavioral changes and net neural effects, and to identify and define the neural mechanisms related to neurobehavioral improvements by providing 30 active or placebo rTMS sessions.

DETAILED DESCRIPTION:
The specific aims (SA) of the CDMRP study are:

SA-1: To determine presence, direction and sustainability of rTMS induced neurobehavioral effects using the DRS (lower scores indicate more function).

SA-2: To determine presence, direction and sustainability of rTMS-induced changes in functional neural activation and whether these changes correlate with improving neurobehavioral function.

SA-3: To determine the rTMS effect on white fiber tracts and whether rTMS-related effects correlate with neurobehavioral gains. White fiber tracts will be examined according to changes in Fractional Anisotropy (FA), Mean Diffusivity (MD), Radial Diffusivity (RD), and Axial Diffusivity (AD).

SA-4: To confirm rTMS safety for severe TBI. The investigators hypothesize that there will be no difference between active and placebo groups according to average number of research related adverse events (AE) during treatment.

To accomplish these aims, the investigators will conduct a double blind, randomized, placebo controlled clinical trial where 58 persons remaining in states of disordered consciousness for 3 to 24 months after TBI are randomized to the active rTMS group or the placebo rTMS group.

The primary outcome is neurobehavioral recovery slope as measured by the total Disability Rating Scale (DRS), which will be collected at bedside at Baseline, Midpoint (15th rTMS Session) and Endpoint (30th rTMS Session). The DRS-PI will be collected weekly via telephone interview for the three weeks between Endpoint and Follow up (3 weeks after 30th rTMS session). Secondary outcomes include four measures of functional neural activation: task related functional magnetic resonance imaging (fMRI), functional connectivity MRI (fcMRI), EEG-Rest and EEG-Task. The functional neural activation measures will be collected at baseline, endpoint and follow up. Motor Threshold Testing and Neurobehavioral measures in addition to the DRS and physical measures will also be collected as secondary outcomes. Motor Threshold testing, neurobehavioral and physical measures will be collected at baseline, midpoint, endpoint and follow up. The additional Neurobehavioral and physical measures are the Disorders of Consciousness Scale-25 (DOCS-25), Coma Recovery Scale Revised (CRS-R), Coma Near Coma Scale (CNC), Modified Tardieu Scale, Modified Ashworth Scale, Spaulding Limb Movement Protocol and the Consciousness Screening Algorithm.

ELIGIBILITY:
Inclusion Criteria:

* At study screening, persons have remained in states of Seriously Impaired Consciousness (SIC) for at least 3 and up to 24 months after TBI
* 18 years of age or older
* Traumatic Brain Injury etiology
* Able to participate in all phases of study including follow-up re-admission
* Able to identify legally authorized representative/surrogate who is able to read and understand informed consent document and provide written consent

Exclusion Criteria:

* Primary injury is a non-traumatic brain injury (and is not secondary to TBI) (e.g., inflammatory, infectious, toxic and metabolic encephalopathies, anoxia, cancer, ischemic and hemorrhagic stroke)
* History of TBI, psychiatric illness (DSM criteria) and or organic brain syndrome (e.g. Alzheimer's)
* Left dorsal lateral pre-frontal cortex (DLPFC) is not accessible (e.g., left frontal lobectomy)
* Incurred large cortically based ischemic infarction subsequent to TBI (size is determined collectively by neurosurgeon, neurologist, neuroradiologist and principal investigator)
* At study screening, patient is receiving anti-epileptic medications to control active seizures
* Have had a documented seizure within 3 months of study screening
* Are ventilator dependent at time of study screening
* Have recovered full consciousness at time of study screening as indicated by a Motor Function scale score of 6 and/or a Communication scale score of 2 on the CRS-R
* Receiving central nervous system (CNS) stimulants that cannot be safely discontinued via titration
* Patient did not speak English prior to injury (bedside testing is conducted in English)
* Pregnant
* Have implanted cardiac pacemaker or defibrillator, cochlear implant or nerve stimulator
* Have MRI or TMS contraindications such as pre-injury claustrophobia, metal in eyes/face or brain
* Other medical conditions, that in investigator's opinion, would preclude subject from completing study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Disability Rating Scale | Change from Baseline in DRS total score at an average 22 days
  The DRS consists of 8 items that address: arousability, awareness and responsivity; cognitive ability for self-care; dependence on others; and psychosocial adaptability. Scores on the DRS range from 0 to 29 with higher scores indicating greater levels of disability.

SECONDARY OUTCOMES:
Disorders of Consciousness Scale-25 | Change from Baseline in DOCS-25 score at 7 days, 14 days, 21 days, 28 days and 50 days
  Neurobehavioral measure that evaluates the subject's responses to sounds, touch, objects, people, tastes, movements and smells
Coma Near Coma Scale | Change from Baseline in CNC total score at an average 22 days
  Neurobehavioral measure that evaluates the subject's responses to sounds, touch, objects, people, tastes, movements and smells
Coma Recovery Scale-Revised | Change from Baseline in CRS-R total score at an average 22 days
  Neurobehavioral measure that evaluates the subject's responses to sounds, touch, objects, people, tastes, movements and smells
Modified Tardieu Scale | Change from Baseline in Modified Tardieu total score at an average 22 days
  Spasticity measure for the following muscles: shoulder flexion, elbow flexion/extension, wrist flexion/extension, hip flexion/extension, knee flexion/extension and ankle extension. The scoring is based on 3 velocities of movement where the higher the rating, the higher degree of muscle tone.
Modified Ashworth Scale | Change from Baseline in Modified Ashworth total score at an average 22 days
  Spasticity measure for the following muscles: shoulder flexion, elbow flexion/extension, wrist flexion/extension, hip flexion/extension, knee flexion/extension and ankle extension. The individual muscle scores will be compared between time points. The higher the rating on the Modified Ashworth the greater degree of muscle tone demonstrated during testing.
Spaulding Limb Movement Protocol | Change from Baseline in Spaudling Limb Movement total score at an average 22 days
  Measures limb movement in response to execution of motor commands in response to 1-step commands that engage upper extremity movements with and without object use.
Consciousness Screening Algorithm | Change from Baseline in consciousness level at 7 days, 14 days, 21 days, 28 days and 50 days
Functional Neuroimaging | Change from Baseline in amount of activation and connectivity at an average 22 days
  Activation in response to a task, resting state and diffusion tensor imaging
EEG Power Spectrum | Change Baseline in EEG frequency power at an average 22 days

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Pape, DrPH, MA, Principal Investigator — Edward Hines Jr. VA Hospital
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Edward Hines, Jr. VA Hospital, Hines, Illinois